CLINICAL TRIAL: NCT03997305
Title: AltaValve Early Feasibility Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 4C Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1890
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency; Mitral Valve Incompetence; Mitral Valve Regurgitation; Mitral Incompetence
Keywords: Mitral Regurgitation; TMVR; Functional Regurgitation; Degenerative Regurgitation; Transcathether Mitral Valve Replacement; Primary Regurgitation; Secondary Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: AltaValve — Transcatheter Mitral Valve Replacement

SUMMARY:
Prospective, single-arm, multicenter study to evaluate the safety and performance of the AltaValve for the treatment of moderate to severe or severe mitral valve regurgitation in subjects who are considered high risk for mortality and morbidity from conventional open-heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years of age.
2. Subjects symptomatic New York Heart Association (NYHA) II-IV.
3. Subjects with severe MR as documented by echo.
4. Subjects who are at high risk for open-heart surgery as documented by the health care professional (e.g., Heart Team consisting of cardiac surgeon and interventional cardiologist in United States).

Abbreviated Exclusion Criteria:

1. Inability to understand the study or a history of non-compliance with medical advice.
2. Unwilling or unable to sign the Informed Consent Form (ICF).
3. History of any cognitive or mental health status that would interfere with study participation.
4. Currently enrolled in any other pre-approval investigational study (does not apply to long-term post-market studies unless these studies might clinically interfere with the current study endpoints (e.g., limit use of study-required medication, etc.)).
5. Female subjects who are pregnant or planning to become pregnant within the study period.
6. Known hypersensitivity or contraindication to aspirin, heparin, or Warfarin without adequate alternative medications.
7. Known hypersensitivity to nitinol (i.e., nickel allergy) that cannot be adequately medicated.
8. Known hypersensitivity to contrast media that cannot be adequately medicated.
9. Evidence of current Left Ventricular Ejection Fraction (LVEF) ≤30% (where current is defined as the latest LVEF measurement completed within 90 days prior to the index procedure).
10. Concurrent medical condition with a life expectancy of less than 12 months.
11. Prior mitral valve repair/replacement (excluding prior surgical mitral valve repair, annuloplasty, or MitraClip not interfering with AltaValve placement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event | 30 days
  Cardiac death, stroke, mitral valve related repeated intervention

SECONDARY OUTCOMES:
Technical success | Index procedure completion (Day 0)
  Technical Success per MVARC criteria
Procedural success | 30 days
  Device success and absence of major device or procedure related serious adverse events
Device success | 30 days
  Device Success per MVARC criteria
Change in MR grade | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Genereux, MD, Principal Investigator — Morristown Medical Center; Vinayak Bapat, MD, Principal Investigator — Allina Health System
Locations (12):
- United States (12):
  - Tucson Medical Center, Tucson, Arizona
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - MedStar Washington Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Morristown Medical Center, Morristown, New Jersey
  - Atrium Health, Charlotte, North Carolina
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Baptist Memorial Hospital - Memphis, Memphis, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott & White, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genereux P, Wrobel K, Ninios V, Grygier M, Tahirkheli N, Sorajja P, Rinaldi MJ, Reardon MJ, Zembala MO, Bezerra HG, Waggoner TE, Giustino G, Waksman R, Grayburn P, Bapat V. 6-Month Outcomes of a Supra-Annular Transcatheter Mitral Valve Replacement: An Early Feasibility Study. JACC Cardiovasc Interv. 2025 Nov 10;18(21):2584-2592. doi: 10.1016/j.jcin.2025.08.040. PMID 41224388